CLINICAL TRIAL: NCT05982678
Title: Basket Study for Oligo-metastatic Breast Cancer Part 1: Trastuzumab-deruxtecan for HER2-positive Oligo-metastatic Breast Cancer
Brief Title: Basket Study for Oligo-metastatic Breast Cancer
Acronym: ANISE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Daiichi Sankyo (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M22BOL
Record Dates: First submitted 2023-07-25; First posted 2023-08-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: HER2-positive Breast Cancer
Keywords: Oligometastatic disease (max 3 lesions)
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab-deruxtecan (Experimental): 5.4mg/kg on a three weekly (21 day) basis, with the goal of 16 cycles leading to a treatment period of year, including local treatment. The first 8 cycles of T-DXd are administered neo-adjuvant, and 8 cycles adjuvant, after completion of local treatment.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — T-DXd 5.4mg/kg on a three weekly (21 day) basis, with the goal of 16 cycles leading to a treatment period of year, including local treatment. The first 8 cycles of T-DXd are administered neo-adjuvant, and 8 cycles adjuvant, after completion of local treatment.

SUMMARY:
The study will include patients with HER2-positive breast cancer and 1- 3 distant metastatic lesions, all amenable for curative intervention. Patients will be stratified by prior therapy and ER expression. In the initial baskets patients with be treated with trastuzumab-deruxtecan.

Patients are treated with T-DXd 5.4mg/kg on a three weekly (21 day) basis, with the goal of 16 cycles leading to a treatment period of year, including local treatment. The first 8 cycles of T-DXd are administered neo-adjuvant, and 8 cycles adjuvant, after completion of local treatment.

The proposed M22BOL trial is based on an important knowledge gap for regarding breast cancer patients with 'oligo-metastatic' disease who are usually not included in clinical trials for patients with metastatic disease since loco-regional treatments (radiation, surgery) with curative intent is not allowed in clinical trials for metastatic breast cancer. Moreover, neo-adjuvant trial protocols for early breast cancer exclude patients with distant metastases that can be treated with curative intent. This basket trial evaluates T-DXd for oligo-metastatic breast cancer with the goal to induce deep responses and subsequently long-lasting disease remissions and potentially cure.

DETAILED DESCRIPTION:
The study will include patients with HER2-positive breast cancer and 1- 3 distant metastatic lesions, all amenable for curative intervention. Patients will be stratified by prior therapy and ER expression. Given the basket-design of this trial other baskets for oligo-metastatic breast cancer can be added, such as but not limited to other breast cancer subtypes or with other promising drugs.

Baskets for de novo oligo-metastatic disease I. ER+/HER2+ II. ER-/HER2+ Baskets for oligo-metastatic disease after prior chemo/anti-HER2 therapy for primary disease III. ER+/HER2+ IV. ER-/HER2+

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of infiltrating HER2-positive breast cancer (as determined by IHC 3+ and/or amplification by ISH)[8]
* Histologic or cytologic proof of breast cancer metastases (at least one lesion)
* Histologic determination of level of ER-expression
* Oligo-metastatic disease as determined by standard of care diagnostics. The number of total individual distant metastases is limited to five, either in one organ or in 2-5 organ systems. Clustered lymph nodes that can be irradiated with curative intent in a single field are defined as single lesion. Pleuritis carcinomatosa, miliary spread of metastases (even within one organ), or peritoneal spread of metastases rules out oligo-metastatic disease and is not allowed. Initial staging by PET-CT (whole body) and MRI of breast and brain are mandatory, as is MRI liver or spine and pelvis in case of liver or bone metastases respectively.
* In case of recurrent disease, a disease-free interval of 24 months.
* Measurable disease according to RECIST1.1
* Patients must be at least 18 years of age and be able to give written informed consent and comply with study procedures.
* World Health Organization (WHO) performance status 0 or 1

Exclusion Criteria:

* prior line of therapy for metastatic disease. Exceptions are endocrine therapy or radiation considered to be part of the curative treatment, within 3 months before enrolment
* leptomeningeal disease or central nervous metastases
* clinically relevant obstruction or compression of spinal cord, central nervous, gastro-intestinal or cardiovascular system, that cannot be alleviated before start of treatment.
* other malignancy, unless treated with curative intention and a long-term survival probability of >95%, including in-situ or pre-malignant lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete radiologic response | up to one year after start treatment
  Number of patients to achieve radiologic response as defined by RECIST 11 with clearnace of ctDNA

SECONDARY OUTCOMES:
Number of patients free of progression | assessed up to 10 years
  as defined by RECIST
Overall Survival | assessed up to 10 years
  time from start treatment to death from any cause
Number of patients with pathological complete response | assessed immediately after surgery
  after resection of primary tumor and/or metastatic lesions after neo-adjuvant treatment
Number of patients with metabolic response | assessed up to 12 months
  as measured with PDG-PET
Number of patients with metabolic response | assessed up to 10 years
  as measured by clearance of ctDNA
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | assessed up to 30 days after last treatment
  determined accoriding to CTCAE v5.0 or Clavien-Dindo (in case of surgical resection)

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Kok, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
to de decided